CLINICAL TRIAL: NCT06068413
Title: A Retrospective, Multicenter, Multiple-viewer-multiple-case (MRMC) Clinical Trial to Evaluate the Safety and Efficacy of CT Image-assisted Detection Software for Focal Liver Lesions
Brief Title: CT Image-assisted Detection Software for Focal Liver Lesions
Acronym: MRMC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Ningbo No.2 Hospital (Other); Shenzhen Sixth People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2023-066
Record Dates: First submitted 2023-09-28; First posted 2023-10-05 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2023-04

CONDITIONS: Focal Liver Lesion
Keywords: CT image-assisted detection software; focal liver lesion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AI-assisted diagnosis (Experimental): Doctors diagnose the focal liver lesion with the help of AI.
  Interventions: Device: CT image-assisted detection software
- common diagnosis (No Intervention): Doctors diagnose the focal liver lesion without the help of AI.

INTERVENTIONS:
Device: CT image-assisted detection software — CT image-assisted detection software can help doctor to diagnosis the focal liver lesion
  Arms: AI-assisted diagnosis

SUMMARY:
To evaluate the safety and effectiveness of the developed and produced CT image-assisted detection software for focal liver lesions before being put into the market.

ELIGIBILITY:
Inclusion Criteria:

* doctors have liver CT scanning experience more than 1 year;

Exclusion Criteria:

* persons don't have the license of practicing physician; doctors don't have liver CT scanning experience or have liver CT scanning experience less than 1 year;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
AFROC | 1 year
  Under different confidence scores, the number of accurately located lesions/the number of true lesions determined by the reference standard was taken as the ordinate coordinate, and (1- the number of negative cases determined by the reference standard/the total number of true negative cases diagnosed by the reference standard) was plotted as the horizontal coordinate

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China